CLINICAL TRIAL: NCT05857839
Title: Effects of Myofascial Release With and Without Support Belt for Sacroiliac Joint Pain, Activity and Disability in Pregnant Females
Brief Title: Myofascial Release With and Without Support Belt for Sacroiliac Joint Pain in Pregnant Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0528
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Sacroiliac Joint Pain
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release with support belt (Experimental): Group A get myofascial release on sacroiliac joint area for up to 600 seconds and total treatment sessions will be 12 in 4 weeks with support belt and a support belt should not be worn for longer than two to three hours at a time and it will be used 4 times a week.
  Interventions: Other: Myofascial release; Other: pelvic Support belt
- Myofascial release without support belt: (Active Comparator): Group B get myofascial release technique to sacroiliac joint area for up to 600 seconds and total treatment sessions will be 12 in 4 weeks but without support belt. Data will be collected and analyzed at baseline and at 4 weeks follow up.
  Interventions: Other: Myofascial release

INTERVENTIONS:
Other: Myofascial release — Patients will get myofascial release technique to sacroiliac joint area for up to 600 seconds and total treatment sessions will be 12 in 4 weeks
Other: pelvic Support belt — The support belt will be worn for less than two to three hours at a time and it will be used 4 times a week
  Arms: Myofascial release with support belt

SUMMARY:
This study will be a randomized controlled trial that will include myofascial release interventions with and without a support belt. 34 Patients will be randomly divided into 2 groups. Assessment will be done by using Numeric Pain Rating Scale, Quebec scale for functional disability, and Pelvic girdle pain questionnaire (PGQ).

DETAILED DESCRIPTION:
Sacroiliac joint dysfunction is a particularly common source of pain during pregnancy and is often an undiagnosed cause of low back pain. In this study, the effects of myofascial release with and without a support belt for sacroiliac joint pain and activity in pregnant females will be analyzed.

Group A of 17 patients will get a myofascial release technique for up to 600 seconds and total treatment sessions will be 12 in 4 weeks with a support belt a support belt should not be worn for longer than two to three hours at a time and it will be used 4 times a week. Group B of 17 patients will also get a myofascial release technique for up to 600 seconds and total treatment sessions will be 12 in 4 weeks but without a support belt. Data will be collected and analyzed at baseline and at 4 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years.
* 2nd and 3rd trimesters of pregnancy.
* The diagnosis of SIJ pain based on tenderness localized to the posterior inferior iliac spine bilaterally with provocative maneuvers of the SIJ in posterior pelvic pain provocation/thigh thrust test, compression test, Gaenslen's test and Patrick's Faber test eliciting considerable pain.
* Positive results from at least three of those provocative tests signified the presence of SIJ pain.

Exclusion Criteria:

* History of rheumatic disease.
* Lumbar spine disc herniation or back injury.
* Previous lumbar spine surgery.
* High risk pregnancy.
* Any bony or soft tissue systemic disease.
* Malignancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 4 weeks
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Quebec scale for functional disability | up to 4 weeks
  The degree of functional disability was estimated using the Quebec scale, assessing 20 routine daily activities on a scale from 0 to 5 (0 = performing activities without difficulty, 1 = performing activities with minimal difficulty, 2 = performing activities with some difficulty, 3 = performing activities with moderate difficulties, 4 = performing activities with greater difficulty, 5 = inability to perform activities). The minimum score was 20 and the maximum score was 100. Higher scores correlate with greater disability.
Pelvic girdle pain questionnaire (PGQ) | up to 4 weeks
  The Pelvic Girdle Questionnaire (PGQ) was also applied. It was created to assess quality of life in patients with pelvic girdle pain during pregnancy and postpartum. It includes 25 questions, with 20 questions aiming to assess activity and 5 questions examining symptoms. Each question is scored on a 4-point Likert type scale (from 'no problem at all' [0 points] to 'to a large extent' [3 points]). The raw scores are then converted into a final score ranging from 0 to 100 (from best to worst outcomes). The questionnaire's reliability and validity in Turkish have been confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Shabbir, MS*, Principal Investigator — Riphah International University
Locations (1):
- Shaikh Zayed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Z, Wu J, Wang X, Wu J, Ren Z. The effects of myofascial release technique for patients with low back pain: A systematic review and meta-analysis. Complement Ther Med. 2021 Jun;59:102737. doi: 10.1016/j.ctim.2021.102737. Epub 2021 May 10. PMID 33984499
- [Background] Laslett M. Evidence-based diagnosis and treatment of the painful sacroiliac joint. J Man Manip Ther. 2008;16(3):142-52. doi: 10.1179/jmt.2008.16.3.142. PMID 19119403
- [Background] Castro-Sanchez AM, Gil-Martinez E, Fernandez-Sanchez M, Lara-Palomo IC, Nastasia I, de Los Angeles Querol-Zaldivar M, Aguilar-Ferrandiz ME. Manipulative therapy of sacral torsion versus myofascial release in patients clinically diagnosed posterior pelvic pain: a consort compliant randomized controlled trial. Spine J. 2021 Nov;21(11):1890-1899. doi: 10.1016/j.spinee.2021.05.002. Epub 2021 May 13. PMID 33991702
- [Background] Mens JM, Damen L, Snijders CJ, Stam HJ. The mechanical effect of a pelvic belt in patients with pregnancy-related pelvic pain. Clin Biomech (Bristol). 2006 Feb;21(2):122-7. doi: 10.1016/j.clinbiomech.2005.08.016. Epub 2005 Oct 7. PMID 16214275
- [Background] Arguisuelas MD, Lison JF, Sanchez-Zuriaga D, Martinez-Hurtado I, Domenech-Fernandez J. Effects of Myofascial Release in Nonspecific Chronic Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2017 May 1;42(9):627-634. doi: 10.1097/BRS.0000000000001897. PMID 28441294
- [Background] Bhat P V, Patel VD, Eapen C, Shenoy M, Milanese S. Myofascial release versus Mulligan sustained natural apophyseal glides' immediate and short-term effects on pain, function, and mobility in non-specific low back pain. PeerJ. 2021 Mar 15;9:e10706. doi: 10.7717/peerj.10706. eCollection 2021. PMID 33777508
- [Background] Elden H, Ladfors L, Olsen MF, Ostgaard HC, Hagberg H. Effects of acupuncture and stabilising exercises as adjunct to standard treatment in pregnant women with pelvic girdle pain: randomised single blind controlled trial. BMJ. 2005 Apr 2;330(7494):761. doi: 10.1136/bmj.38397.507014.E0. Epub 2005 Mar 18. PMID 15778231